CLINICAL TRIAL: NCT03339830
Title: European Registry of Patients With Infantile-onset Spinal Muscular Atrophy
Status: Completed | Type: Observational
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Other Study IDs: IO-SMA-Registry; 2017-A02291-52 (Other: ANSM (French Regulatory Authority))
Record Dates: First submitted 2017-10-18; First posted 2017-11-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Spinal Muscular Atrophy
Keywords: SMA; Spinal Muscular Atrophy; Neuromuscular disease; Spinraza
MeSH Terms: conditions — Muscular Atrophy, Spinal; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
IO-SMA-Registry is a prospective, longitudinal and observational study which objective is to collect prospectively information on longevity, psychomotor development and respiratory function of patients with infantile-onset spinal muscular atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Muscular Atrophy diagnosed in childhood (before 18 months) and genetically confirmed.
* For patients with SMA type 1: Never acquired independent sitting position (more than 30 seconds, without hand support or any external support)
* For patients with SMA type 2 or 3: Patient treated with a market approved treatment for SMA or with a treatment in an expanded access program
* Any age
* Patients over 18 years of age or parent(s)/legal guardian(s) of patients < 18 years of age not opposed to data collection for research purposes

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neuromuscular reference centers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in survival | Baseline and then every 6 months until the end of the study, up to 5 years
Change from Baseline in psychomotor development | Baseline and then every 6 months until the end of the study, up to 5 years
  Motor milestones acquired and/or lost
Change from Baseline in the number of lower track infections | Baseline and then every 6 months until the end of the study, up to 5 years
Change from Baseline in ventilation use | Baseline and then every 6 months until the end of the study, up to 5 years
Change from Baseline in cough assist use | Baseline and then every 6 months until the end of the study, up to 5 years
Change from Baseline in Forced Vital Capacity | Baseline and then every 6 months until the end of the study, up to 5 years
Change from Baseline in diurnal saturation | Baseline and then every 6 months until the end of the study, up to 5 years
Change from Baseline in nocturnal hypercapnia | Baseline and then every 6 months until the end of the study, up to 5 years

SECONDARY OUTCOMES:
Change from the beginning of the treatment of psychomotor development | Since the beginning of the treatment until the end of the study, up to 5 years
  Retrospective and prospective collection of data from patients/parents interview and medical files Motor milestones acquired and/or lost
Change from the beginning of the treatment of the number of hospitalizations | Since the beginning of the treatment until the end of the study, up to 5 years
  Retrospective and prospective collection of data from patients/parents interview and medical files
Change from the beginning of the treatment of the duration of hospitalizations | Since the beginning of the treatment until the end of the study, up to 5 years
  Retrospective and prospective collection of data from patients/parents interview and medical files
Change from Baseline of Clinical Global Impressions - Improvement (CGI-I) | Baseline and then every 6 months until the end of the study, up to 5 years
  Quantification of patient progress and treatment response over time
Change from Baseline of the scoliosis occurence | Baseline and then every 6 months until the end of the study, up to 5 years
Change from Baseline of the arthrodesis occurence | Baseline and then every 6 months until the end of the study, up to 5 years
Change from Baseline of contractures occurrence | Baseline and then every 6 months until the end of the study, up to 5 years
Change from Baseline of wheelchair use | Baseline and then every 6 months until the end of the study, up to 5 years
Change from Baseline of feeding status | Baseline and then every 6 months until the end of the study, up to 5 years
  Feeding difficulties (swallowing, chewing, sucking), excessive drooling, need of a feeding tube, occurrence of gastrostomy
Change from Baseline of speech impairment | Baseline and then every 6 months until the end of the study, up to 5 years
  Speech incapacity, voice tone disorders
Change from Baseline of Hammersmith Infant Neurological Examination (HINE) score | Baseline and then every 6 months until the end of the study, up to 5 years
Change from Baseline of Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP-INTEND) score | Baseline and then every 6 months until the end of the study, up to 5 years
Change from Baseline of Motor Function Measure (MFM) score | Baseline and then every 6 months until the end of the study, up to 5 years
Change from Baseline of Expanded Hammersmith Functional Motor Scale (HFMSE) score | Baseline and then every 6 months until the end of the study, up to 5 years
Change from Baseline of the number of physiotherapy sessions per week | Baseline and then every 6 months until the end of the study, up to 5 years
Change from Baseline of the number of balneotherapy sessions per week | Baseline and then every 6 months until the end of the study, up to 5 years
Change from Baseline of the number of occupational therapy sessions per week | Baseline and then every 6 months until the end of the study, up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Servais, MD, PhD, Principal Investigator — Institute of Myology
Locations (6):
- France (6):
  - Hopital Morvan - CHU de Brest, Brest
  - Service de Rééducation Pédiatrique Infantile " L'Escale " - Hôpital Femme Mère Enfant, Bron
  - Hôpital le Bocage - CHU Dijon, Dijon
  - Maladie Neuromusculaire de l'enfant - Service Maladies infectieuses et neurologie infantile - Hôpital Roger Salengro, Lille
  - I-Motion Institute, Paris
  - Unité de neurologie pédiatrique - Hôpital des enfants, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided